CLINICAL TRIAL: NCT06982664
Title: Effect of Preserving the Left Colic Artery on Proximal Bowel and Anastomotic Blood Perfusion During Radical Resection for Rectal Cancer: A Randomized Controlled Trial Based on Laser Speckle Contrast Imaging
Brief Title: Effect of Preserving the Left Colic Artery on Proximal Bowel Perfusion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo Medical Center Lihuili Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KY2025PJ104
Record Dates: First submitted 2025-04-16; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Rectal Cancer Surgery; Perfusion Imaging; Anastomosis, Leaking
Keywords: rectal caner; Perfusion; Anastomosis leakage; Laser Speckle Contrast Imaging

STUDY DESIGN:
Intervention Model Description: Patients were categorized into two groups, HT and LT, based on the planned management of the IMA.
  HT Group: In the HT group, the IMA was ligated approximately 1 cm from its origin after meticulous dissection of the surrounding tissue to ensure clear visualization of the IMA root.
  LT Group: In the LT group, the surgical approach focused on preserving the LCA. Apical lymph node dissection was performed around the origin of the IMA. The superior rectal artery was ligated distal to the origin of the LCA.
  As part of the prospective cohort sub-study in the LT group, the preserved LCA underwent temporary, controlled occlusion intraoperatively. This was done after confirming LCA preservation and before colonic transection or anastomosis. The aim was to assess perfusion changes-such as retraction of the ischemic demarcation line using LSCI-to evaluate the functional role of the LCA. After assessment, the occlusion was released to restore blood flow.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study employs single-blinding where patients are unaware of their treatment allocation (High Tie [HT] or Low Tie [LT]). The operating surgeon is necessarily unblinded intraoperatively to perform the assigned surgical technique. The statistician(s) performing the data analysis will be masked to treatment group assignments until the analysis is complete. Randomization is managed by a designated investigator using pre-generated random numbers after eligibility confirmation (1:1 ratio to HT or LT group).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HT Group (Experimental): In this group, the IMA was ligated approximately 1 cm from its origin. With this approach, both the LCA and the inferior mesenteric vein were ligated near the lower border of the pancreas.
  Interventions: Procedure: High Tie of Inferior Mesenteric Artery
- LT Group (Experimental): In the LT group, apical lymph node dissection was performed around the origin of the IMA. During this procedure, the LCA was identified and preserved and the superior rectal artery was ligated.
  Interventions: Procedure: Low Tie of Inferior Mesenteric Artery

INTERVENTIONS:
Procedure: High Tie of Inferior Mesenteric Artery — IMA was ligated approximately 1 cm from its origin after dissection of the surrounding tissue to ensure clear visualization of the IMA root. Using this technique, the LCA and the inferior mesenteric vein were ligated near the lower border of the pancreas
  Arms: HT Group
Procedure: Low Tie of Inferior Mesenteric Artery — During this procedure, the LCA was identified and preserved, and the superior rectal artery was ligated. Before colonic transection or anastomosis, the preserved LCA underwent temporary, controlled occlusion. After assessing perfusion changes using LSCI, the occlusion was released to restore blood flow.
  Arms: LT Group

SUMMARY:
Patients with rectal or rectosigmoid cancer undergoing radical resection will be randomly assigned to either high-tie (HT) or low-tie (LT) ligation of the Inferior Mesenteric Artery (IMA). Proximal bowel blood perfusion will be measured using Laser Speckle Contrast Imaging, and the perfusion characteristics will be compared between the two ligation groups.

Additionally, for participants randomized to the LT group, an embedded prospective cohort sub-study will be performed. This sub-study involves controlled, temporary intraoperative occlusion of the preserved Left Colic Artery (LCA). During this temporary occlusion, LSCI will be used to assess the resulting changes in colonic perfusion, specifically measuring outcomes like the ischemic demarcation line (LOD) retraction distance, to further investigate the functional contribution of the preserved LCA. The overall trial aims to determine the optimal IMA ligation strategy based on objective perfusion data and a deeper understanding of LCA's role.

DETAILED DESCRIPTION:
The primary goal of this clinical trial is to compare proximal bowel blood perfusion following HT versus LT of the IMA during anterior resection for rectal cancer. LSCI will be used to assess perfusion in both groups.Additionally, this trial incorporates an embedded prospective cohort sub-study, which will be conducted specifically within the LT group, where the Left Colic Artery (LCA) is preserved. The purpose of this sub-study is to further elucidate the impact of this LCA preservation on left colonic perfusion in these patients. This will be achieved by investigating the retraction distance of the ischemic demarcation line following temporary occlusion of the preserved LCA under LSCI guidance, and by exploring potential anatomical and pathophysiological factors that may contribute to variations in this retraction distance.

The main questions the study seeks to answer are:

Does HT ligation result in significantly different proximal bowel blood perfusion, as measured by LSCI, compared to LT ligation? Does knowledge of intraoperative bowel perfusion, as assessed by LSCI, influence surgical decision-making, specifically regarding changes to the planned transection line? Are there significant differences in quantified perfusion intensity at the transection line between HT and LT ligation techniques? What is the retraction distance of the ischemic demarcation line, observed via LSCI, following temporary occlusion of the LCA, and what are the potential anatomical or pathophysiological factors associated with variations in this distance? Patients undergoing anterior resection for rectal cancer will be randomized to receive either HT or LT ligation of the IMA. LSCI will be used intraoperatively to assess bowel perfusion.

Participants will:

Undergo anterior resection for either rectal or rectosigmoid cancer, with HT or LT ligation of the IMA determined by the randomization process.

Have bowel perfusion assessed intraoperatively using LSCI. Have the maximum perfusion distance (MPD) measured as the primary outcome for the main randomized trial component.

Have the perfusion intensity at the transection line quantified as a secondary outcome.

Have any changes to the planned transection line documented based on intraoperative LSCI findings, as a secondary outcome.

As part of the embedded prospective cohort sub-study, undergo temporary intraoperative occlusion of the LCA with subsequent LSCI assessment to measure the retraction distance of the ischemic demarcation line.

As part of the embedded prospective cohort sub-study, have data collected on relevant potential anatomical (e.g., vascular anatomy variations) and pathophysiological factors (e.g., presence of atherosclerosis, patient comorbidities) that may influence the ischemic demarcation line retraction distance.

This trial aims to provide high-level evidence to inform and optimize IMA management strategies during anterior resection for rectal or rectosigmoid cancer, based on proximal bowel perfusion assessment using LSCI visualization, and to provide deeper mechanistic insights into the specific role and functional importance of the LCA in maintaining colonic perfusion.

ELIGIBILITY:
Inclusion Criteria:

1. a confirmed diagnosis based on pathological reports;
2. patients who had not received any prior treatment;

Exclusion Criteria:

1. a history of previous abdominal surgery or neoadjuvant chemotherapy/radiation affecting bowel perfusion or anastomosis;
2. patients requiring emergency surgery due to acute complications;
3. intraoperative findings necessitating a shift to alternative procedures, such as local excision, abdominoperineal resection, Hartmann's operation, or intersphincteric resection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Perfusion Distance (MPD) | Perioperative
  Determined by measuring the distance from the ischemic line of demarcation to the starting point of the sigmoid colon.

SECONDARY OUTCOMES:
Number of participants requiring revision of the planned bowel transection line following intraoperative Laser Speckle Contrast Imaging (LSCI)-based bowel perfusion assessment | Perioperative
  This measure quantifies the number of participants whose planned bowel transection line, initially determined by conventional intraoperative assessment (e.g., visual inspection, serosal sheen, peristalsis, mesenteric pulse palpation), is revised after LSCI is used to assess bowel perfusion. Revisions occur under two conditions:
  1. The initial transection line was planned distal to the Line of Demarcation (LOD) indicated by LSCI, and the surgeon adjusts the transection line based on the LSCI findings (typically moving it proximally).
  2. The initial transection line was planned proximal to the LSCI-indicated LOD, but the surgeon determines it must be moved distally to ensure a tension-free anastomosis.
  If the initial transection line is proximal to the LSCI LOD and bowel length is sufficient for a tension-free anastomosis, no revision is counted. Data will be reported as the total count and percentage of participants who meet the revision criteria.
Speckle Flow Index (SFI) at the Proximal Anastomosis Site Measured by Laser Speckle Contrast Imaging (LSCI) | Perioperative
  This measure reports the microvascular blood perfusion at the planned proximal bowel anastomosis site, assessed intraoperatively using Laser Speckle Contrast Imaging (LSCI) and SIM BFI Software (V2.0). The metric used is the Speckle Flow Index (SFI), a numerical value calculated by the software.
  The SFI quantifies the relative speed of red blood cells in the tissue, derived from 50 consecutive image frames with a 10 ms exposure time. While LSCI also generates real-time 2D perfusion maps for visual guidance, this measure focuses on the SFI value alone.
  The SFI is reported as a numerical value, typically in arbitrary perfusion units (APU) or relative units. Statistical analysis will summarize these SFI values across participants, reporting measures such as mean, median, and standard deviation.
Ischemic Demarcation Line (LOD) Retraction Distance | Perioperative
  This outcome measure will be assessed exclusively in participants randomized to the LT group. Before temporarily occluding the preserved LCA, the initial LOD will be identified using LSCI and marked. Then, the LCA will be temporarily occluded using a non-damaging vascular clamp. LSCI will be used again to visualize colonic perfusion and identify the new LOD. The LOD retraction distance is defined as the proximal distance along the bowel from the previously established reference point to the new LOD identified via LSCI. This measurement will be recorded in centimeters (cm).

OTHER OUTCOMES:
Intraoperative blood loss | Perioperative
  Total blood lost during surgery, calculated as suctioned volume plus gauze weight change, recorded in milliliters (ml).
Operative time | Perioperative
  Duration of the surgical procedure, from skin incision to wound closure, recorded in minutes.
Intraoperative blood transfusion | Perioperative
  Occurrence of blood transfusion during surgery, recorded as Yes/No.
Postoperative surgical complications | Perioperative
  Graded using the Clavien-Dindo classification system from the end of surgery until hospital discharge.
Anastomotic leakage rate | Perioperative
  Anastomosis leakage is diagnosed by triple contrast CT in case of suspected ananstomosis leakage. Additionally colonoscopy may be performed. Anastomosis severity is graded as follows: local infection without abscess, abscess without clear intraluminal bowel connection, abscess with intraluminal bowel connection, free perforation to abdominal cavity.
Length of hospital stay | Perioperative
  Number of days from the day of surgery to the day of hospital discharge, recorded in days.

CONTACTS AND LOCATIONS:
Overall Officials: Jiazi Yu, M.D., Study Director — Ningbo Medical Center of Lihuili Hospital

IPD SHARING:
Plan to Share IPD: Yes
All data generated in this study will be made available in the main publication or its supplementary materials. Additional de-identified datasets will be shared upon reasonable request from qualified researchers after completion of the study and approval by the institutional ethics committee.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Individual participant data (IPD) and supporting documents will be available beginning 6 months after publication of the study results and will remain available for a period of 3 years.
Access Criteria: Qualified researchers affiliated with academic institutions, hospitals, or research organizations may request access to the de-identified individual participant data (IPD), study protocol, and statistical analysis plan. Data will be shared for research purposes only, following submission and approval of a research proposal and data access agreement.